CLINICAL TRIAL: NCT03187665
Title: The Ties That Bind: Evaluation of a Patient-worn Pulse Oximeter Compared to Traditional Pulse Oximetry on Loss of Signal Integrity in Pediatric Patients
Brief Title: Alarms Due to Loss of Signal Integrity in Partially Wireless Versus Traditional Pulse Oximetry in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Pamela Petersen (Other)
Responsible Party: Sponsor-Investigator, Pamela Petersen, Pediatric Critical Care Fellow, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Other Study IDs: 953341-1
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: Pediatric; Pulse Oximeter; Wireless; Motion; False Alarm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- 1-6 years: 12 subjects in the age range of 1-6 years old.
  Interventions: Device: Radical 7; Device: Radius 7
- 6-10 years: 12 subjects in the age range of 6-10 years old.
  Interventions: Device: Radical 7; Device: Radius 7
- 11-17 years: 12 subjects in the age range of 11-17 years old.
  Interventions: Device: Radical 7; Device: Radius 7

INTERVENTIONS:
Device: Radical 7 — The Radical 7 is the traditional wall-connected pulse oximeter currently used at Children's Hospital of Wisconsin (CHW) which requires a 12 foot cable connecting the patient to a wall unit. While being continuously monitored with the Radical 7 pulse oximeter, subjects will be asked to complete age appropriate activities. The pulse oximetry data will be analyzed for instances of alarm state corresponding to loss of signal integrity as defined by complete inability to pick up the subject signal or a change in the pulse oximetry saturation value by 4%.
  Other Names: Masimo Radical 7 Pulse Oximeter
Device: Radius 7 — The Radius 7 is a newer, partially wireless pulse oximeter which eliminates the cable connecting the patient to a wall unit by instead connecting to a small device worn on the patient's arm or leg. The small device then sends the continuous pulse oximeter data wirelessly to the central monitoring station. While being continuously monitored with the Radius 7 pulse oximeter, subjects will be asked to complete age appropriate activities. The pulse oximetry data will be analyzed for instances of alarm state corresponding to loss of signal integrity as defined by complete inability to pick up the subject signal or a change in the pulse oximetry saturation value by 4%.
  Other Names: Masimo Radius 7 Pulse Oximeter

SUMMARY:
This research study will help the investigators to learn more about a device used when children are sick called a pulse oximeter. The pulse oximeter measures how much oxygen is inside a child's blood without taking blood from the child. It is non-invasive meaning it does not enter the body. The device has a cable attached to it. At the end of the cable is a wrap that looks like a Band-Aid with a red light on it. This wrap is placed around a finger or toe. The red light gives the investigators a reading of how much oxygen is in the child's blood and the child's heart rate. Having a pulse oximeter connected to a child is painless. This device is used in many places. Besides hospitals, it is used in doctors' offices and in fitness centers.

This study will help the investigators learn more about whether a partially wireless, more portable pulse oximeter that connects to a small device worn on the child's arm or leg will give the investigators a more reliable signal/reading while letting children move more easily. The investigators will compare this device with the traditional wall-connected unit. Movement of the cable or a child moving may give a false oxygen reading. The investigators will ask the child to do activities that create movement and will look at the readings when the child moves. The investigators think the partially wireless pulse oximeter will be more reliable during movement than the traditional wall-connected unit.

Subjects will have two continuous pulse oximeter probes placed on them. These soft probes will go on a finger, toe, foot or hand and will be attached to two different pulse oximeter monitors. The child will then be asked to do common childhood activities based on their age for about 20 minutes. These activities will be play activities the child already does such as grabbing a toy, drawing with crayons or kicking a ball. Continuous pulse oximetry data will be recorded during the testing and will be stored in a way that it cannot be linked to the subject after the testing is complete.

DETAILED DESCRIPTION:
PURPOSE OF THE STUDY This study will evaluate the loss of signal integrity secondary to motion in pediatric subjects being monitored with a newer, partially wireless pulse oximeter (the Radius 7) which eliminates the cable connecting the subject to a wall unit by instead connecting to a small device worn on the subject's arm or leg. The Radius 7 will be compared to the traditional wall-connected pulse oximeter currently used at Children's Hospital of Wisconsin (CHW) which requires a cable connecting to a wall unit (the Radical 7).

HYPOTHESIS Continuously monitoring pulse oximetry with a partially wireless monitor without physical connection to a wall unit will decrease episodes of loss of signal integrity generated by motion artifact in healthy pediatric subjects completing age appropriate activities.

BACKGROUND, SIGNIFICANCE, AND RATIONALE Pulse oximetry is used in both inpatient and outpatient environments to measure the oxygen saturation in a person's blood and the pulse, or heart rate. Pulse oximeters use a painless Band-Aid-like probe that attaches to a fingertip, toe, hand or foot and shines a light through the skin. The monitor then determines how much oxygen is in the blood and the pulse rate based on the way the light passes through the skin. The probe is connected to the monitor by a cable of varying lengths. Movement can cause incorrect pulse oximeter measurements.

Continuous pulse oximetry is considered a standard of care in pediatric intensive care units; however pediatric patients have a high incidence of false alarms in part due to motion artifact. These false alarms contribute to the 94% false alarm incidence in pediatric ICU patients. (Lawless) Motion artifact is potentially exacerbated by the long cables connecting the patients to the continuous monitors. Currently the FDA has not approved any completely cable-free pulse oximeters for continuous use; however Masimo has produced a device (the Radius 7) that overcomes the previously required cable connection to a wall unit via wireless transmission from a patient-worn continuous monitor. (Masimo) There are currently no studies looking at this patient worn monitor in relation to the motion artifacts that frequently cause false alarms in pediatric patients.

The Joint Commission has listed alarm fatigue as a top patient safety concern and as of January 1, 2016 has required hospitals to establish policies and procedures for managing alarm fatigue. Reduction in false alarms is necessary to reduce alarm fatigue. This pilot study will use clinical data to measure the effect of eliminating this cable-to-wall connection on motion artifact. Additionally, early mobility in critically ill patients has been shown to improve outcomes. Freeing patients from one of the cables currently tying them to the room may decrease the false alarms from motion artifact while simultaneously improving mobility, therefore improving patient outcomes and safety.

DESIGN AND METHODS Subjects: Healthy pediatric subjects ranging from 6 months to 17 years of age. Pediatric subjects will be recruited via fliers placed in pediatric critical care areas, in the Translational Research Control Unit (TRU) and on the MCW research bulletin board outside the MCW office of research. Subjects may include those responding to the fliers directly as well as the healthy siblings of patients being evaluated or treated in the Children's Hospital of Wisconsin Emergency Room (EDTC), Clinics or Hospital.

Setting: The Children's Hospital of Wisconsin (CHW): primarily in the TRU designed to mimic a CHW outpatient clinic room; and also including available sites near the EDTC or clinic to facilitate making testing more convenient for the subject's family if the subject is a healthy sibling of a patient being evaluated in the EDTC or clinic.

Procedures:

While being continuously monitored on the current equipment used by CHW (the wall-connected Radical 7) and the partially wireless Radius 7 pulse oximeter, subjects will be asked to complete age appropriate activities as developed by CHW physical therapists, for approximately twenty minutes. These activities include common childhood activities such as kicking a ball or drawing with crayons. If a subject declines to participate in an activity, an alternate will be suggested. The investigators will analyze the pulse oximetry data for instances of alarm state corresponding to loss of signal integrity as defined by complete inability to pick up the subject signal or a change in the pulse oximetry saturation value by 4%. (Seixas, Seixas and Pereira)

Endpoints: Enrollment of and data acquisition on 48 pediatric subjects: 12 in each of the following developmental age groups: 6 month-1year, 1-6 years, 6-10 years, and 11-17 years.

Data analysis:

All data will be collected in a de-identified manner in which subjects will be given a study case number and all data will be collected under that case number.

The number of episodes of loss of signal integrity leading to an alarm state generated by the wall-connected Radical 7 unit compared to the partially wireless Radius 7 unit during completion of the developmentally appropriate activities will be compared. Analysis will be performed by the Quantitative Health Sciences department at MCW and a 20% reduction in episodes of loss of signal integrity will be considered clinically significant.

TOTAL NUMBER OF HUMAN RESEARCH PARTICIPANTS PROPOSED FOR THIS STUDY. 48 pediatric subjects: 12 in each of the following developmental age groups: 6 months-1year, 1-6 years, 6-10 years, and 11-17 years. This number of participants will provide representative data for a pilot study investigating the most common age groups seen in the pediatric ICU in order to identify the age groups most likely to benefit from further study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between the ages of 6 months and 17 years at the time of data acquisition.

Exclusion Criteria:

* Subjects will be excluded if they have any pre-existing cardiac or pulmonary chronic medical diagnoses as determined by asking the subject's guardian.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The subjects will be a sampling from the communities served by the Children's Hospital of Wisconsin. Pediatric subjects will be recruited via fliers placed in pediatric critical care areas, in the Translational Research Control Unit (TRU) and on the Medical College of Wisconsin (MCW) research bulletin board outside the MCW office of research. Subjects may include those responding to the fliers directly as well as the healthy siblings of patients being evaluated or treated in the Children's Hospital of Wisconsin Emergency Room (EDTC), Clinics or Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
instances of alarm state corresponding to loss of signal integrity | 20 minutes
  Loss of signal integrity is defined as complete inability to pick up the patient signal or a change in the pulse oximetry saturation value by 4%.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela C Petersen, M.D., Principal Investigator — Medical College of Wisconsin Affiliated Hospitals, Inc.; Sheila Hanson, M.D., Principal Investigator — Medical College of Wisconsin Affiliated Hospitals, Inc.
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, Masimo, who makes both of the pulse oximeters, will be able to see de-identified information. They will not be allowed to see "Protected Health Information" (PHI). IPD that will be shared includes Subject Number, Age, Race, Gender, Probe Location (dominant vs. nondominant hand), Activity (Likert score), Start time of activity, Stop time of activity, Radius 7 Probe location, Radical 7 Probe location, Instance of alarm state Radius 7, Duration of alarm state Radius 7, Loss of signal integrity Radius 7-Change in pulse ox saturation of 4% or more, Loss of signal integrity Radius 7-no signal, Instance of alarm state Radical 7, Duration of alarm state Radical 7, Loss of signal integrity Radical 7-Change in pulse ox saturation of 4% or more, and Loss of signal integrity Radical 7-no signal. This de-identified data with no PHI will be shared via USB stick or e-mail electronically.

REFERENCES:
- [Background] Lawless ST. Crying wolf: false alarms in a pediatric intensive care unit. Crit Care Med. 1994 Jun;22(6):981-5. PMID 8205831
- [Background] Seixas DM, Seixas DM, Pereira MC, Moreira MM, Paschoal IA. Oxygen desaturation in healthy subjects undergoing the incremental shuttle walk test. J Bras Pneumol. 2013 Jun-Aug;39(4):440-6. doi: 10.1590/S1806-37132013000400007. PMID 24068265